CLINICAL TRIAL: NCT02238340
Title: Oxycodone Extended-release in the Treatment of Perioperative Pain in Patients Undergoing Orthopaedic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Central Dr. Luis Ortega (Other)
Responsible Party: Principal Investigator, Beatriz Arismendi Gómez, Medico Anestesiologo, Hospital Central Dr. Luis Ortega
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Oxycodone
Record Dates: First submitted 2014-09-02; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Surgery
Keywords: Postoperatory pain; Oxycodone
MeSH Terms: interventions — Ketoprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Extended-release oxycodone 10mgr (Experimental): Extended-release oxycodone 10 mgrs , started 12 hours before orthopaedic surgery
  Interventions: Drug: Extended-release oxycodone; Drug: Extended- release Oxycodone; Drug: ketoprofen; Drug: dipirone; Drug: dexametasone; Drug: Morphine IV (rescue)
- Extended-release oxycodone 20 mgr (Experimental): Extended-release oxycodone 20 mgr , started 12 hours before orthopaedic surgery
  Interventions: Drug: Extended-release oxycodone; Drug: Extended- release Oxycodone; Drug: ketoprofen; Drug: dipirone; Drug: dexametasone; Drug: Morphine IV (rescue)

INTERVENTIONS:
Drug: Extended-release oxycodone — 10 o 20 mgrs of extended-release oxycodone ,started 12 hours before orthopaedic surgery
Drug: Extended- release Oxycodone
Drug: ketoprofen
  Other Names: Both groups received ketoprofen
Drug: dipirone
  Other Names: Both groups received dipirone
Drug: dexametasone
  Other Names: Both groups received dexametasone
Drug: Morphine IV (rescue)
  Other Names: Both groups received Morphine IV (rescue)

SUMMARY:
Inadequate control of acute postoperative pain (DAPO) brings deleterious consequences for the patient, including significant cardiovascular and respiratory complications. Apart from the human suffering that is undeniable pain. Schemes oral analgesia with opioids for the treatment of DAPO, have shown to be as or more effective than intravenous or epidural regimes, and less expensive. Comparing the effectiveness of 10 to 20 mgs of oxycodone sustained release for 12 hours before surgery, into two groups of 20 patients (O-10, O-20) undergoing orthopedic surgery, in a scheme involving multimodal ketoprofen, dipyrone metoclopramide and dexamethasone. Values were recorded visual analog scale (VAS)for pain at rest and effort, requirement for rescue intravenous morphine and incidence of side effects to the entry and exit of the PACU (T0, TE) and at 6 and 18 hours postoperatively (T6, T18),and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients between 18 and 60 years old, both sexes, undergoing elective orthopedic surgery.

Exclusion Criteria:

* Use of psychotropic medication or illicit drug use
* Pregnancy
* Liver disease
* Opioid use
* History of postoperative nausea and vomiting
* Ileus
* Allergy or intolerance to any of the study drugs
* Physical or mental inability to use the pain scale, or any surgical complications.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Percents of patients with EVA < 4 to the alt of UCPA, and 6 , 18 postoperatory hours | 24 hours

SECONDARY OUTCOMES:
Percents of patients with adverse events because of treatment | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz S Arismendi Gomez, MD, Principal Investigator — Sociedad Venezolana de Anestesiologia
Locations (1):
- Servicio de Aestesiologia.Hospital "Dr Luis Ortega", Porlamar, Nueva Esparta, Venezuela